CLINICAL TRIAL: NCT00739687
Title: A Double-Blind, Placebo-Controlled, Randomized Trial Evaluating the Efficacy and Safety of Alagebrium (ALT-711) in Patients With Chronic Heart Failure
Brief Title: Safety & Efficacy of ALT-711 (Alagebrium) in Chronic Heart Failure
Acronym: BENEFICIAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been termination early due to financial constraints.
Sponsor: Synvista Therapeutics, Inc (Industry)
Responsible Party: Adriaan A. Voors, MD, PhD, University Medical Center Groningen, Groningen, The Netherlands
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-711-0527a
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure
MeSH Terms: interventions — alagebrium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALT-711 (Experimental): Alagebrium 200 mg BID
  Interventions: Drug: ALT-711
- Placebo (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALT-711 — 200 mg tablet BID for 9 months.
  Other Names: Alagebrium
  Arms: ALT-711
Drug: Placebo — 200 mg tablet BID for 9 months.
  Arms: Placebo

SUMMARY:
Several lines of evidence have suggested that Advanced Glycation End-products (AGEs) play a role in the development and progression of heart failure. The AGE-crosslink breaker Alagebrium improved cardiac function and symptoms in experimental preclinical and small human heart failure studies. These results have not yet been confirmed in a randomized controlled clinical trial. Objective: to evaluate the safety and efficacy of alagebrium in subjects diagnosed with heart failure. This is a randomized, double-blind, placebo-controlled trial to assess the effects of 400 mg (2 x 100 mg bid) of alagebrium versus placebo over 9 months. 100 subjects will be studied (50 per treatment group) in approximately 6 centers. Procedures: exercise testing (VO2 max; the primary variable), ECGs and blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* NYHA II-IV heart failure
* Echocardiographic ejection fraction ≤ 45% (echo does not need to be repeated at the screening visit if a prior echo is on record which indicates an ejection fraction < 40%)
* Duration of heart failure > 3 months
* Stable heart failure medical therapy for > 1 month
* Patients need to be able to understand content of and willing to provide informed consent

Exclusion Criteria:

* Patient ≤ 18 years
* History of myocardial infarction in previous 6 months
* History of stroke/TIA/RIND in previous 6 months
* Severe valvular dysfunction
* Severe pulmonary disease
* History of systemic inflammatory or collagen vascular disease
* Active and or treated malignancies within 12 months prior to inclusion
* Any significant condition either medical or non-medical that could lead to difficulty complying with the protocol
* Patients on cardiac resynchronisation therapy (CRT) or scheduled for CRT implantation
* Pacemaker therapy (unless rescue pacing at ≤ 40 bpm) or scheduled pacemaker implantation
* History of valve replacement or surgery
* Uncontrolled diabetes mellitus (HbA1c > 9.5%)
* Clinically significant renal disturbance (sMDRD calculated GFR≤30 mL/min/1.73m2; sMDRD is calculated as 186 x serum Cr (mg/dl)-1.154 x years-0.203 x (0.742 if female) x (1.210 if African American)
* Clinically significant liver disease (ASAT/ALAT > 2,5 times the upper limit of normal)
* Severe anemia at baseline (Hemoglobin <10 g/dl or <6.2 mmol/l)
* Use of any investigational drug(s) within 30 days prior to screening
* Pregnancy or active breast-feeding (urine pregnancy tests will be performed on all female subjects of childbearing potential)*
* Active pericarditis/myocarditis
* The inability of patients to undergo exercise testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
The primary end-point of the study will be aerobic capacity (VO2 max) measured at exercise testing. An improvement of 15% in VO2 max will be considered as a clinically significant increase. | 9 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama Hospital, Birmingham, Alabama
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina